CLINICAL TRIAL: NCT02130674
Title: Improvement of Therapy in Patients With Severe Traumatic Brain Injury: Differential Impact of Local and Systemic Changes and Routinely Applied Drugs
Brief Title: Optimized Therapy in Severe Traumatic Brain Injured Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Fresenius Kabi (Industry); University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, John Stover, Prof. Dr. med., University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNF 111782; SNF 111782 (Other Grant/Funding Number: SNF 111782)
Record Dates: First submitted 2014-04-26; First posted 2014-05-05 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Traumatic Brain Injury; Coma
Keywords: traumatic brain injury; glutamine; microdialysis; metabolism
MeSH Terms: conditions — Brain Injuries, Traumatic; Coma | interventions — alanylglutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dipeptiven (Experimental): 0.75 g/ kg/ d Dipeptiven ( L- alanine- L- glutamine; 82 mg/ ml L- alanine, 134.6 mg/ ml L- glutamine; Fresenius Kabi, Switzerland) continuous intravenous infusion
  Interventions: Drug: Dipeptiven

INTERVENTIONS:
Drug: Dipeptiven — two groups: group 1: continuous infusion for 24 hours group 2: continuous infusion for 5 days
  Other Names: Dipeptamin

SUMMARY:
Severe traumatic brain injury is associated with life-threatening and incapacitating secondary injury.

Contemporary therapeutic interventions are aimed at preventing and treating secondary damage. In this context, improved cerebral metabolism is an important target in modern neurointensive care.

The main hypothesis is that continuous intravenous infusion of glutamyl-alanyl dipeptide restores disturbed brain metabolism following severe traumatic brain injury.

DETAILED DESCRIPTION:
Patients suffering from severe traumatic brain injury and requiring multimodal neuromonitoring during pharmacological coma will receive alanyl-glutamine dipeptide (Dipeptiven) as part of standard clinical nutrition.

In two groups of patients the influence of different duration of infusion (group 1: 24 hours; group 2: 5 days) will be investigated. For this, pharmacokinetic and pharmacodynamic parameters in plasma and brain are determined.

Increased plasma glutamine and alanine in arterial and jugular venous plasma and in cerebral microdialysates are to reflect efficacy of Dipeptiven infusion.

Plasma glutamate levels as well as changes in cerebral glutamate, lactate, lactate/pyruvate ratio, intracranial pressure, bispectral index electroencephalography will be measured to exclude potential adverse effects

ELIGIBILITY:
Inclusion Criteria:

* severe traumatic brain injury
* prolonged pharmacologic coma
* multimodal neuromonitoring (microdialysis, ptiO2)
* enteral nutrition

Exclusion Criteria:

* patients anticipated to decease within 48 hours
* abdominal injury
* mass transfusion
* renal impairment
* hepatic impairment
* barbiturate coma
* parenteral nutrition
* weight below 50 kg
* weight above 100 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
plasma glutamine levels | 2 to 7 days
  changes in plasma glutamine levels during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute (micromole/ liter) or relative (%) values
cerebral glutamine | 2 to 7 days
  changes in cerebral glutamine levels during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute (micromole/ liter) or relative (%) values

SECONDARY OUTCOMES:
cerebral lactate | 2 to 7 days
  changes in cerebral lactate and lactate/pyruvate ratio reflecting cerebral energetic deficit during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute (millimole/ liter) or relative (%) values
cerebral lactate to pyruvate ratio | 2 to 7 days
  changes in lactate/pyruvate ratio reflecting cerebral energetic deficit during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute (millimole/ liter) or relative (%) values
cerebral glutamate | 2 to 7 days
  changes in cerebral glutamate reflecting cerebral energetic deficit during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute (micromole/ liter) or relative (%) values
intracranial pressure | 2 to 7 days
  changes in intracranial pressure reflecting brain edema during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute (mm Hg) or relative (%) values
bispectral index electroencephalography | 2 to 7 days
  changes in bispectral index EEG reflecting neuronal activation during and after infusion of alanyl-glutamine compared to baseline and intra-infusion values expressed in absolute or relative (%) values

CONTACTS AND LOCATIONS:
Overall Officials: John F Stover, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Nageli M, Fasshauer M, Sommerfeld J, Fendel A, Brandi G, Stover JF. Prolonged continuous intravenous infusion of the dipeptide L-alanine- L-glutamine significantly increases plasma glutamine and alanine without elevating brain glutamate in patients with severe traumatic brain injury. Crit Care. 2014 Jul 2;18(4):R139. doi: 10.1186/cc13962. PMID 24992948